CLINICAL TRIAL: NCT05266651
Title: Efficiency of Tadalafil for Management of Female Sexual Dysfunction in Females With Genital Mutilation
Brief Title: Efficiency of Tadalafil for Management of Female Sexual Dysfunction
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Hussein Aly Hussein, Assistant professor, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22022022
Record Dates: First submitted 2022-02-22; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Sexual Dysfunction
Keywords: female genital mutilation; Sexual dysfunction; Clitoral artery Doppler
MeSH Terms: conditions — Sexual Dysfunction, Physiological | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tadalafil group (Active Comparator): 5 mg of Tadalafil on daily bases for one month duration
  Interventions: Drug: Tadalafil 5mg
- placebo group (Placebo Comparator): the patients will receive oral tablets without any active substance for one month
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tadalafil 5mg — oral tablets for one month duration
  Arms: tadalafil group
Drug: Placebo — oral tablets for one month duration
  Arms: placebo group

SUMMARY:
comparative study between tadalafil versus placebo effect for the management of circumsized female

DETAILED DESCRIPTION:
the group of patient will be randomly divided into 2 groups, half of the patients will receive tadalafil and the other half will receive placebo

ELIGIBILITY:
Inclusion Criteria:

* female with history of female genital mutilation female with history of sexual dysfunction

Exclusion Criteria:

* any medical disorder

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-03-10 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
clitorial Artery Doppler | after one month duration of drug use
  Pulsatile index
Clitorial artery doppler | after one month duration of drug use
  Resistance index
Clitorial artery doppler | after one month duration of drug use
  Peak systolic velosity

SECONDARY OUTCOMES:
score of sexual function | after on month of the drug use
  arousal orgasm frequency

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Elainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
the exel sheet
Supporting Information: Study Protocol, SAP